CLINICAL TRIAL: NCT04743817
Title: Feasibility Evaluation of the OtoSet - Ear Cleaning System
Brief Title: Feasibility Evaluation of OtoSet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SafKan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SK-0119
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Cerumen Impaction of Both Ears

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- OtoSet - Ear Cleaning Sytem (Experimental)
  Interventions: Device: OtoSet - Ear Cleaning System

INTERVENTIONS:
Device: OtoSet - Ear Cleaning System — Up to five (5) cleaning cycles using the OtoSet - Ear Cleaning System

SUMMARY:
This is a single center study. 100 ears are planned (up to 100 patients). Each subject will have one or both ears cleaned with OtoSet. The subject's level of earwax will be evaluated before and after by an evaluator.

DETAILED DESCRIPTION:
This is a single center study. 100 ears are planned (up to 100 patients). Each subject will have one or both ears cleaned with OtoSet. The subject's level of earwax will be evaluated before and after by an evaluator.

Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

Total duration of subject participation will be 1 day with a follow up call within 2-4 days after the procedure. Total duration of the study is expected to be 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Mild (1), Moderate (2), or Complete (3) occlusion of the ear canal based on the Degree of Occlusion Scale in one or both ears
* Informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient of the quality of data
* Subject has life threatening illness
* Subject has immune deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Efficacy as Assessed by Occlusion Scale | Treatment Visit (Day 1) (pre- to post-procedure)
  Improvement of 1.0 on the Degree of Occlusion Scale (4 point scale) pre- and post-procedure evaluation (score 0 = no occlusion; 3 = complete occlusion)
Safety as Assessed by Adverse Events | Treatment Visit (Day 1) through follow-up call (Day 2-4)
  Incidence of adverse events with severity defined using the National Cancer Institute's Common Terminology Criteria for Adverse Events (4 point scale) (1 = mild; 4 = life-threatening)

CONTACTS AND LOCATIONS:
Overall Officials: Felice Anderson, Principal Investigator — Eclipse Clinical Research; Ronald Brazg, MD, FACE, Principal Investigator — Rainier Clinical Research Center
Locations (2):
- United States (2):
  - Eclipse Clinical Research, Tucson, Arizona
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No